CLINICAL TRIAL: NCT00985387
Title: Persistence of Solifenacin Treatment in Overactive Bladder Patients in Real Life Practice: A 12-month, Prospective, Multicenter, Open-label, Observational Study
Brief Title: Evaluation of Adherence to Solifenacin Treatment in Overactive Bladder Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPK-1
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Urinary Bladder, Overactive; Overactive Bladder
Keywords: Solifenacin; Overactive bladder; persistency of the treatment; Vesicare
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solifenacin treatment: Male and female OAB patients who were treated with solifenacin
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — oral
  Other Names: YM905; Vesicare

SUMMARY:
The purpose of the study is to assess patient's persistency in maintaining solifenacin treatment for overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder symptoms lasting for more than 3 months
* The question 3 score of the overactive bladder symptom score(OABSS)≥ 2 and the sum score of OABSS ≥ 3
* Symptoms of urinary urgency defined as a level of 1 to 2 in a 3-point Urgency Perception Scale (UPS)

Exclusion Criteria:

* Any condition that would contraindicate their usage of anticholinergic treatment, including: urinary retention, gastric retention, uncontrolled narrow angle glaucoma, myasthenia gravis
* Symptomatic acute urinary tract infection (UTI)
* Diagnosed or suspected of interstitial cystitis
* Treatment with anticholinergic drugs for over 3 months within 12 months prior to the study
* Pregnant or nursing women
* Treatment within the 14 days before the study or expected to initiate treatment during the study with any anticholinergic drugs other than solifenacin or treatment for overactive bladder with other drugs
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OAB patients who were treated with solifenacin
Sampling Method: Non-Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
percentage of patients who are maintaining solifenacin treatment | Month 0, Month 1, Month 3, Month 6, Month 9 and Month 12

SECONDARY OUTCOMES:
percentage of patients who discontinued solifenacin treatment | Month 0, Month 1, Month 3, Month 6, Month 9 and Month 12
percentage of patients who switched to other OAB medication | Month 0, Month 1, Month 3, Month 6, Month 9 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (18):
- South Korea (18):
  - Bucheon-si
  - Busan
  - Chuncheon
  - Daegu
  - Daejeon
  - Gangneung
  - Gumi
  - Gwangju
  - Gyongju
  - Hwasun
  - Iksan
  - Inchon
  - Jeonju
  - Masan
  - Seongnam
  - Seoul
  - Suwon
  - Ulsan